CLINICAL TRIAL: NCT07179432
Title: Effectiveness of Facial Mask Non-Invasive Ventilation in Adults Under General Anesthesia: Two-Hand C-E vs V-E Techniques. A Double-Blind Randomized Trial
Brief Title: Effectiveness of Facial Mask NIV in Adults Under General Anesthesia: Two-Hand C-E vs V-E Techniques
Acronym: VENTMASK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Mario Zamudio, University professor with a master's degree in clinical epidemiology, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IN31-2024
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: General Anesthetics
Keywords: ventilation; mask ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial with two parallel groups, randomized 1:1, superiority design, blinded to the patient and data analyst.
Who Masked: Participant, Outcomes Assessor
Masking Description: Generation of the Random Allocation Sequence The sequence will be generated using the latest version of R software with permuted blocks of 2, 4, and 6 participants with variable block sizes, and one stratification variable: use of an oropharyngeal cannula.
  Allocation Concealment Mechanism The allocation will be kept in an opaque envelope that does not allow the assigned group to be seen.
  Implementation The envelope will be opened only by one of the investigators after completing the inclusion criteria and signing the informed consent
  Blinding Patient: Will be blinded as they will be under general anesthesia Outcome Evaluator Will be blinded as their analysis will be conducted on videos recorded by the research team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-Hand V-E Maneuver Facial Mask Ventilation. (Experimental): The V-E maneuver is achieved by placing the thumbs and thenar eminence of each hand on the sides of the mask, creating a "V" shape, while the rest of the fingers perform a jaw thrust described as an "E" shape. This will be performed after anesthetic induction when the patient is unconscious and apneic.
  Interventions: Procedure: V-E facial mask ventilation maneuver
- C-E facial mask ventilation maneuver (Active Comparator): The C-E maneuver is achieved by placing the thumb and index finger of each hand on the mask in a "C" shape, while the third, fourth, and fifth fingers of both hands perform a jaw thrust towards the mask in an "E" shape. This will also be performed after anesthetic induction when the patient is unconscious and apneic.
  Interventions: Procedure: C-E facial mask ventilation maneuver

INTERVENTIONS:
Procedure: V-E facial mask ventilation maneuver — The V-E maneuver is achieved by placing the thumbs and thenar eminence of each hand on the sides of the mask, creating a "V" shape, while the rest of the fingers perform a jaw thrust described as an "E" shape. This will be performed after anesthetic induction when the patient is unconscious and apneic. The C-E maneuver is achieved by placing the thumb and index finger of each hand on the mask in a "C" shape, while the third, fourth, and fifth fingers of both hands perform a jaw thrust towards the mask in an "E" shape. This will also be performed after anesthetic induction when the patient is unconscious and apneic.
  Arms: Two-Hand V-E Maneuver Facial Mask Ventilation.
Procedure: C-E facial mask ventilation maneuver — The C-E maneuver is achieved by placing the thumb and index finger of each hand on the mask in a "C" shape, while the third, fourth, and fifth fingers of both hands perform a jaw thrust towards the mask in an "E" shape. This will also be performed after anesthetic induction when the patient is unconscious and apneic.
  Arms: C-E facial mask ventilation maneuver

SUMMARY:
This study aims to compare two different ways doctors hold a face mask to help the participant breathe during general anesthesia. The investigators are evaluating which method, the "C-E" or the "V-E" technique, works best.

If the participant chooses to take part, on the day of surgery, after anesthesia has been administered and the participant is asleep, the doctor will use one of these two mask-holding techniques to assist breathing for a short period. The investigators will measure how effectively the participant is breathing, check carbon dioxide levels, and record the doctors' assessment of how easy and comfortable each technique was for them. This study will not alter any other aspect of the surgery or recovery.

DETAILED DESCRIPTION:
Airway management is a routine part of an anesthesiologist's work when subjecting patients to different degrees of sedation, eventually reaching general anesthesia. It is also crucial in emergency care, where general practitioners, emergency physicians, and prehospital care technicians/technologists (APH) manage the airway, each with varying degrees of training and experience. In these scenarios, the doctor or APH provider will determine whether to maintain the airway using invasive or non-invasive methods to achieve proper ventilation. Factors such as patient characteristics, which may predict difficult mask ventilation combined with difficult laryngoscopy, include: Mallampati classification III or IV, obesity (BMI over 30 kg/m²), presence of teeth, history of obstructive sleep apnea, short thyromental distance, limited mandibular protrusion, cervical mass, limited neck extension, presence of a beard, male gender, or age over 46 years.

However, it has been observed that predictions about difficult mask ventilation or difficult intubation only correspond to actual difficult airway scenarios 25% of the time. Furthermore, difficult intubation and difficult mask ventilation were unanticipated in 93% and 94% of cases, respectively. Other factors that influence patient outcomes include the patient's current condition based on the context, such as elective surgery versus an emergency scenario. This can be the same patient at two different times, but the approach may vary depending on the physician's training and experience, whether it is an APH technician/technologist, a general practitioner, an emergency physician, or an anesthesiologist. These decisions are also influenced by the availability of equipment.

Mask ventilation is often considered intuitive, but it has been demonstrated to be difficult to learn and apply in both hospital and prehospital settings . In such scenarios, the face mask should always be available and serves as the initial approach before invasive airway management or rescue if intubation or a supraglottic device fails. Therefore, proper training in face mask ventilation skills, including the two-hand technique, is necessary to improve the seal, mandibular protrusion, and neck extension, targeting the determinants of difficult mask ventilation as defined by the ASA: "The inability to provide adequate ventilation (e.g., confirmed by detection of end-tidal carbon dioxide) due to any of the following: inadequate mask seal, excessive gas leak, or excessive resistance to gas entry or exit".

For two-handed mask ventilation, two techniques have been described: the C-E technique, in which the thumb and index fingers of each hand form a "C" around the mask while the third, fourth, and fifth fingers pull the jaw towards the mask in an "E" shape, and the V-E technique, in which the thumbs and thenar eminence of each hand press against the sides of the mask in a "V" shape while the rest of the fingers perform the "E" jaw traction .

Current evidence points to better performance of the V-E maneuver compared to the C-E maneuver. However, the performance of these maneuvers has not been uniformly evaluated with the use of adjuncts to face mask ventilation, such as the Guedel airway, or in patients under neuromuscular blockade.

Given the lack of scientific evidence, the results of our research would not only impact the work of anesthesiologists but also extend to emergency services and prehospital settings. This would lead to improved patient outcomes by enhancing knowledge of two-hand mask ventilation and raising the quality of care provided to patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years old
* Scheduled for elective surgery
* Require general anesthesia
* Consent to participate in the study

Exclusion Criteria:

* Presence of predictors of difficult ventilation: presence of a beard, --obstructive sleep apnea/hypopnea syndrome
* Anticipated difficult airway
* Classified as ASA IV or higher
* Oxygen saturation less than 92% upon admission
* Requirement for supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation ml/kg | 10 minutes during procedure
  Average ventilation in milliliters per kilogram of body weight for seven ventilations recorded on the anesthesia machine at the end of expiration.

SECONDARY OUTCOMES:
Average CO2 mmHg | 10 minutes during procedure
  Average CO2 in mmHg for seven ventilations recorded on the anesthesia machine at the end of expiration.
Ineffective ventilation | 10 minutes during procedure
  Proportion of ineffective ventilation, defined as ventilation less than 1.5 ml/kg.
Operator satisfaction. | 10 minutes during procedure
  Operator's perceived ease of use, on a Likert scale from 1 to 5, with 1 being very easy and 5 being very difficult.
Hypoxemia | 10 minutes during procedure
  defined as SpO2 less than 92%

OTHER OUTCOMES:
Adverse events by group. | Perioperative/Periprocedural
  Adverse events by group.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Zamudio, Anesthesiologist, Principal Investigator — Universidad de Antioquia
Locations (2):
- Colombia (2):
  - Hospital alma Mater de Antioquia, Medellín, Antioquia
  - Antioquia´s University, Medellín

IPD SHARING:
Plan to Share IPD: Yes
by contact to the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at least five years
Access Criteria: contact to investigator

REFERENCES:
- [Background] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Kovacs G, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Jones PM; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 2. Planning and implementing safe management of the patient with an anticipated difficult airway. Can J Anaesth. 2021 Sep;68(9):1405-1436. doi: 10.1007/s12630-021-02008-z. Epub 2021 Jun 8. PMID 34105065
- [Background] Kheterpal S, Han R, Tremper KK, Shanks A, Tait AR, O'Reilly M, Ludwig TA. Incidence and predictors of difficult and impossible mask ventilation. Anesthesiology. 2006 Nov;105(5):885-91. doi: 10.1097/00000542-200611000-00007. PMID 17065880
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT07179432/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT07179432/ICF_001.pdf